CLINICAL TRIAL: NCT00004040
Title: Patients With Chronic Lymphocytic Leukemia or Multiple Myeloma Whose Disease Has Been Controlled With Chemotherapy: Rituximab Anti-CD20 Monoclonal Antibody or Interferon Alpha 2-b as Maintenance Therapy
Brief Title: Monoclonal Antibody Therapy or Biological Therapy in Treating Patients With Chronic Lymphocytic Leukemia or Multiple Myeloma in Remission After Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patient accruals
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Purpose: Treatment
Other Study IDs: CDR0000066763; CBRG-9806; NCI-V98-1495
Record Dates: First submitted 1999-12-10; First posted 2004-08-05 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Neoplasms, Plasma Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Interferon-alpha; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Biological therapies such as interferon alfa-2b use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase II trial to study the effectiveness of rituximab or interferon alfa-2b in treating patients who have chronic lymphocytic leukemia or multiple myeloma in remission.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of rituximab or interferon alfa-2b maintenance therapy in patients with chronic lymphocytic leukemia or multiple myeloma in remission after chemotherapy. II. Determine the progression free survival, failure free survival, and overall survival of these patients from time of chemotherapy discontinuation to completion of maintenance therapy. III. Compare the survival rates of these patients to similar patients treated in published studies. IV. Determine the quality of life of these patients on these regimens.

OUTLINE: Patients enter one of two treatment arms: Arm I: Patients receive rituximab IV on days 1, 8, 15, and 22 for course 1, and then once a month for 11 months or until disease progression. Arm II: Patients receive subcutaneous interferon alfa-2b every other day three times per week for 12 months. Quality of life is assessed monthly during therapy. Patients are followed every 3 months for 1 year, and then annually for up to 5 years.

PROJECTED ACCRUAL: A total of 60-80 patients (30-40 per disease type) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: B-cell chronic lymphocytic leukemia or multiple myeloma in remission that was previously treated with chemotherapy without disease progression

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Lymphocyte count less than 10,000/mm3 Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception No active infection or other concurrent lifethreatening disease Medical condition satisfactory for treatment with chemotherapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-06; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Cancer Biotherapy Research Group
Locations (3):
- United States (3):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - St. Joseph Regional Cancer Center, Bryan, Texas